CLINICAL TRIAL: NCT00687297
Title: A Randomized Phase II Study Evaluating Vandetanib (ZD6474) in Combination With Docetaxel and Carboplatin Followed by Placebo or Maintenance Therapy With Vandetanib in Patients With IIIb, IV or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Vandetanib Combined With Chemotherapy to Treat Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PrE0501; IRUSZACT0088 (Other: AstraZeneca)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Stage IIIB Non Small Cell Lung Cancer; Stage IV Non Small Cell Lung Cancer; Vandetanib; Docetaxel plus carboplatin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Docetaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vandetanib Maintenance (Active Comparator): Docetaxel day 1, carboplatin day 1 + vandetanib induction days 1 through 21 (daily) of a 28-day cycle for 4 cycles. If free of disease progression after 4 cycles, vandetanib maintenance daily until progression.
  Interventions: Drug: vandetanib induction; Drug: Docetaxel; Drug: Carboplatin; Drug: Vandetanib maintenance
- Placebo Maintenance (Placebo Comparator): Docetaxel day 1, carboplatin day 1 + vandetanib induction days 1 through 21 (daily) of a 28-day cycle for 4 cycles. If free of disease progression after 4 cycles, placebo maintenance daily until progression.
  Interventions: Drug: vandetanib induction; Drug: Docetaxel; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: vandetanib induction — 100 mg daily by mouth
  Other Names: ZD6474
Drug: Docetaxel — (75mg/m2) IV (in the vein) on day 1 of a 21-day cycle for 4 cycles or until disease progression
  Other Names: Taxotere
Drug: Carboplatin — IV (in the vein) to area under the curve (AUC) of 6 on day 1 of a 21 day cycle, for 4 cycles or until disease progression
Drug: Placebo
  Arms: Placebo Maintenance
Drug: Vandetanib maintenance — 300 mg daily by mouth
  Other Names: ZD6474
  Arms: Vandetanib Maintenance

SUMMARY:
It has been shown in previous studies that the ability to treat lung cancer could be significantly improved by not only targeting the tumor cells directly with chemotherapy, but also by cutting off the blood supply to the cancer cells. Blood vessels that supply the tumor are formed through a process called angiogenesis. Vandetanib is an investigational drug that acts by producing what is called an anti-angiogenic effect. An Anti-angiogenic effect is able to inhibit the development of new blood vessels required by tumors to survive by blocking the growth factors needed to form new blood vessels.

The purpose of this study is to determine if the addition of vandetanib to a standard chemotherapy regimen will slow or stop the growth of the cancer for a longer period of time compared to the time period generally gained from the use of standard chemotherapy alone

DETAILED DESCRIPTION:
Lung cancer is the number one cause of cancer-related mortality in the United States, with an estimated 160,390 deaths in 2007. Over 80% of these patients will have non-small cell lung cancer (NSCLC), and the majority of these patients have advanced disease at the time of diagnosis.

Patients with advanced disease who have an adequate performance status clearly benefit from systemic chemotherapy, and many clinical trials have been carried out to determine the most effective regimen. Comorbidities associated with NSCLC preclude the use of cisplatin in doublet therapies, and, a meta-analysis comparing platinum-based doublet regimens to non-platinum based, third generation regimens revealed that survival outcomes between these regimens were equivalent. Despite poor response and overall survival benefits in this patient population with accepted treatment doublets, the addition of a third cytotoxic agent did not improve survival and demonstrated increased toxicity. Therefore, it appears a threshold maximum response can be gained with cytotoxic chemotherapy alone. However, the poor outcomes still associated with advanced NSCLC clearly demanded the need for continued improvements in treatment. It was postulated that anticancer therapy could be significantly improved by not only targeting the tumor cells directly, but also by targeting neo-angiogenesis. A randomized phase II trial demonstrated a significant improvement in time to progression (TTP) in patients receiving carboplatin, paclitaxel and bevacizumab compared to chemotherapy alone. Due to life-threatening and fatal hemorrhage patients with squamous cell histology, as well as those with a prior history of hemoptysis and brain metastases were excluded from all further clinical trials using bevacizumab. The definitive study of bevacizumab in NSCLC was a randomized phase III clinical trial conducted by ECOG (E4599) in which patients with advanced non-squamous NSCLC received carboplatin + paclitaxel with or without bevacizumab which met the clinical endpoint of improvement in survival and led to the approval of bevacizumab in first line treatment in patients with advanced NSCLC with non-squamous histology.

The epidermal growth factor receptor (EGFR) protein activation leads to TK activation and results in cell proliferation, motility, adhesion, invasion, survival, and angiogenesis. The EGFR is over expressed in many solid tumors, including non-small cell lung cancer (NSCLC), and multiple studies have suggested a shortened survival in NSCLC patients whose tumor over expresses EGFR . Although studies using small-molecule TK inhibitors (TKIs) in NSCLC did not meet efficacy endpoints, a phase III trial demonstrated the benefit of EGFR TKI monotherapy. Patients with advanced NSCLC who have received 2 or 3 prior therapies were randomized to erlotinib or placebo, and those receiving erlotinib demonstrated a survival benefit that led to FDA approval of this drug in 2004.

The studies above clearly demonstrated a benefit to combining anti-angiogenic factors with chemotherapy, and as a monotherapy using anti-EGFR agents, in patients with advanced NSCLC. The potential benefit to simultaneously targeting these 2 pathways has been addressed in the recurrent disease setting.

Vandetanib is a novel oral molecule (anilinoquinazoline) that has dual activity against both the VEGFR and EGFR pathways. Specifically, this compound has potent and reversible inhibitory activity against VEGFR-2 (KDR), VEGFR-3 (Flt-4), EGFR and RET . Vandetanib is a TKI and thus acts through inhibition of ATP binding to the tyrosine kinase domains of these receptors. Recombinant enzyme assays have demonstrated that vandetanib is highly selective for both VEGFR-2 (IC50=40 nm) with only slightly lower affinity for VEGFR-3 (2.7 fold). EGFR tyrosine kinase activity is inhibited with an IC50=500 nm. The results of a second-line setting phase II trial were presented by Heymach et al at the ASCO meeting in 2006. In this trial, patients were randomized to receive either docetaxel alone, or docetaxel with either 100mg or 300mg of vandetanib. Patients with squamous cell histology, controlled brain metastases and prior history of hemoptysis were allowed on study. The primary endpoint of prolongation of progression-free survival (PFS) was met in the 100mg arm (Hazard Ratio(HR) 0.64, p=0.07). There was no increased incidence of hemoptysis in patients receiving vandetanib, and no CNS hemorrhage events were observed, and side effects commonly attributed to EGFR inhibition (rash, diarrhea) were higher on the 300mg arm. Early combination studies suggest that in patients with NSCLC, vandetanib is safe in combination with chemotherapy, may improve the outcomes of chemotherapy when used at the 100 mg dose, and has activity as monotherapy at the 300mg dose. In addition, none of the observed hemorrhagic complications seen with bevacizumab were observed, even in patients at high risk for this complication.

In this study, our main goal is to study the combination of docetaxel + carboplatin and vandetanib, followed by a double-blind randomized assignment to maintenance therapy with vandetanib 300 milligrams (mg) or placebo by mouth daily until disease progression to determine if maintenance therapy can prolong progression-free survival. In addition to clinical efficacy outcomes we will monitor for safety and tolerability, as well as explore any differences in outcome based on age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Advanced disease (stage IIIB disease [malignant pleural or pericardial effusion seen on CT or Chest X-ray, any N, M0] or stage IV disease [Any T, any N, M1: distant metastases]) that is primary or recurrent
* Measurable disease according to the RECIST criteria
* ECOG Performance Status 0 or 1
* Adequate organ function, as evidenced by ALL the following
* Absolute neutrophil count (ANC) ≥ 1500/mm³ and platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 gm/dL
* Total bilirubin ≤ 1 X institutional ULN; if patient has Gilbert's disease, then patient must have isolated hyperbilirubinemia (e.g. no other liver function test abnormality), with maximum bilirubin ≤ 2 X institutional ULN.
* AST, ALT and alkaline phosphatase (Alk Phos) must be ≤ 1.5 ULN
* Creatinine ≤ 1.5 X institutional ULN or calculated creatinine clearance ≥ 60 ml/min
* Potassium between 4 mEq/L and institutional ULN (supplementation may be used),
* Calcium (ionized or adjusted for albumin)within institutional normal limits
* Magnesium within institutional normal limits (supplementation may be used)
* No prior cytotoxic chemotherapy or targeted therapy for advanced or metastatic disease (Prior adjuvant therapy for lung cancer allowed if completed > 1 year prior to registration)
* Able to take oral medication

Exclusion Criteria:

* Myocardial infarction, superior vena caval syndrome, NYHA classification of heart disease ≥ 2 within the 3 months prior to entry
* History of an uncontrolled or recurrent ventricular, supraventricular or nodal arrhythmia that requires treatment
* Hypertension not controlled by medication
* Peripheral or sensory neuropathy > grade 1
* Known hypersensitivity to carboplatin or docetaxel
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (30):
- United States (30):
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - SwedishAmerican Hospital, Rockford, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Ochsner Clinic, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - St. Joseph Mercy Hospital- Ann Arbor, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Ocean Medical Center, Brick, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Aultman Hospital, Canton, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hematology & Oncology of NEPA, Dunmore, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central PA Hematology & Medical Oncology Associaties, Lemoyne, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - The Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Sanford Clinic, Sioux Falls, South Dakota
  - Meharry Medical College, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Result] Aisner J, Manola JB, Dakhil SR, Stella PJ, Sovak MA, Schiller JH. Vandetanib plus chemotherapy for induction followed by vandetanib or placebo as maintenance for patients with advanced non-small-cell lung cancer: a randomized phase 2 PrECOG study (PrE0501). J Thorac Oncol. 2013 Aug;8(8):1075-83. doi: 10.1097/JTO.0b013e3182937317. PMID 23689430
- See also: Vandetanib in Advanced Non-Small Cell Lung Cancer — https://www.ncbi.nlm.nih.gov/pubmed/23689430

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized to Vandetanib Maintenance: Docetaxel (75mg/m2)IV (in the vein) + Carboplatin IV (AUC=6) day 1 of 21 day cycle + vandetanib (100mg) days 1 through 21 (daily) x 4 cycles. If SD, PR CR after 4 cycles --> Maintenance treatment: vandetanib (300mg) daily until progression [1 Cycle= 28 days]
- Randomized to Placebo Maintenance: Docetaxel (75mg/m2)IV (in the vein) + Carboplatin IV (AUC=6) day 1 of 21 day cycle + vandetanib (100mg) days 1 through 21 (daily) x 4 cycles. If SD, PR CR after 4 cycles --> Maintenance treatment: Placebo 3 tablets daily until progression [1 Cycle= 28 days]
Period: Randomization
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance
Started | 80 | 82
Completed | 77 | 81
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Withdrew before treatment, ineligible | 1 | 1
Period: Induction
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance
Started | 77 | 81
Completed | 32 | 26
Not Completed | 45 | 55
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Adverse Event | 16 | 15
Not completed — Death | 7 | 11
Not completed — Lack of Efficacy | 17 | 21
Not completed — Ineligible | 0 | 1
Not completed — Patient Noncompliance | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Other | 0 | 1
Period: Maintenance
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance
Started | 32 | 26
Completed | 29 | 25
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Continuous [Median (Full Range); unit: years] | 63.5 [38 to 84] | 63 [36 to 82] | 63 [36 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 42 | 42 | 84
Region of Enrollment [Number; unit: participants]
  United States | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from randomization (prior to induction) to first evidence of disease progression or death without progression. Participants alive without progression were censored at the date of last disease evaluation.
Time Frame: Assessed every 2 cycles (1 cycle = 3 weeks during induction and 4 weeks during maintenance))
Population: All randomized patients were included.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Randomized Patients: All patients enrolled in the study
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 162
Months | 4.5 [3.6 to 4.9]

2. Secondary Outcome: Objective Response Rate
Description: Best overall response (complete or partial response), assessed using RECIST criteria (version 1.0)
Time Frame: Assessed every 2 cycles (1 cycle = 3 weeks during induction and 4 weeks during maintenance))
Population: All randomized patients were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance
Number analyzed (Participants) | 82 | 80
percentage of participants | 18.8 [10.9 to 29.0] | 18.3 [10.6 to 28.4]
Statistical Analysis 1: Comparison: Randomized to Vandetanib Maintenance vs Randomized to Placebo Maintenance; Fisher's exact test with two-sided Type I error of 5% was used to test the null hypothesis of no difference in response rate between arms; Test type: Superiority or Other; p = 1.00, Fisher Exact; Mean Difference (Final Values) = 0.5

3. Secondary Outcome: Progression-free Survival
Description: Time from randomization to first evidence of disease progression or death. Patients alive without progression are censored at the date of last disease evaluation.
Time Frame: every 2 cycles (every 6 weeks during induction, every 8 weeks during maintenance)
Population: All randomized patients were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized to Vandetanib Maintenance | Randomized to Placebo Maintenance
Number analyzed (Participants) | 80 | 82
months | 4.5 [3.3 to 5.8] | 4.2 [2.8 to 4.9]
Statistical Analysis 1: Comparison: Randomized to Vandetanib Maintenance vs Randomized to Placebo Maintenance; There was 80% power to detect a 50% improvement in median progression-free survival, using a stratified log-rank test with one-sided Type I error of 10%; Test type: Superiority or Other; p = 0.02, Regression, Cox — p-value from Wald test; The model was adjusted for gender (male vs. female) and stage (Stage IIIB vs. Stage IV/Recurrent); Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.07 to 2.07]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every 3 weeks during induction and every 4 weeks during maintenance.
Description: Serious adverse events are defined as events of grade 3 or higher that were considered possibly, probably, or definitely treatment-related. Other adverse events include grade 1 or 2 events possibly, probably or definitely treatment-related occurring at a rate of 5% or higher.
Groups:
- Treated on Vandetanib Maintenance: Adverse events among patients receiving Vandetanib using the maintenance phase of the study
- Treated on Placebo Maintenance: Adverse events among patients receiving placebo during the maintenance phase of the study
- All Treated Patients - Induction: Adverse events occurring during induction among all treated patients
Arm/Group | Treated on Vandetanib Maintenance | Treated on Placebo Maintenance | All Treated Patients - Induction
Serious Adverse Events (participants affected / at risk) | 22/32 | 11/26 | 111/157
Other Adverse Events (participants affected / at risk) | 29/32 | 22/26 | 145/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated on Vandetanib Maintenance (N=32) | Treated on Placebo Maintenance (N=26) | All Treated Patients - Induction (N=157)
Allergic Reaction (Immune system disorders) | 0 | 0 | 3
Anorexia (Gastrointestinal disorders) | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 2
Cardiac - other (Cardiac disorders) | 1 | 0 | 1
Colitis, infectious (Gastrointestinal disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 5
Depression (Psychiatric disorders) | 0 | 0 | 1
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 3 | 0 | 14
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Extremity - limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 12
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 10
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 4
Hemorrhage - other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Infection w grade 3-4 neutrophils, lung (Infections and infestations) | 0 | 0 | 3
Infection w/unk ANC, abdomen NOS (Infections and infestations) | 0 | 0 | 1
Infection w/unk ANC, liver (Infections and infestations) | 0 | 0 | 1
Infection w/unk ANC, lung (Infections and infestations) | 0 | 1 | 2
Infection - other (Infections and infestations) | 0 | 0 | 3
Insomnia (General disorders) | 0 | 0 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Leukocytes increased (Blood and lymphatic system disorders) | 0 | 0 | 25
Lung hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lymphopenia (Investigations) | 0 | 0 | 1
Metabolic/Laboratory, other (Metabolism and nutrition disorders) | 0 | 0 | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 0 | 2
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 65
Nonneuropathic generalized weakness (Nervous system disorders) | 0 | 0 | 4
Perforation, colon (Gastrointestinal disorders) | 0 | 0 | 1
Photosensitivity (Eye disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 3
QTc Interval prolonged (Investigations) | 1 | 0 | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 2 | 6
Skin - other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 9
Upper GI hemorrhage, NOS (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Weight loss (Investigations) | 1 | 0 | 1
AST, SGOT Increased (Investigations) | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 0 | 1 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chest/thoracic pain NOS (Reproductive system and breast disorders) | 1 | 2 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Death, disease progression NOS (General disorders) | 2 | 0 | 0
Dental/teeth/periodontal pain (Gastrointestinal disorders) | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
GI - other (Gastrointestinal disorders) | 0 | 1 | 0
Infection w/gr 0-2 neutrophils, lung (Infections and infestations) | 1 | 0 | 0
Infection w/Unk ANC, stomach (Infections and infestations) | 1 | 0 | 0
Neuropathy, motor (Nervous system disorders) | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Taste disturbance (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated on Vandetanib Maintenance (N=32) | Treated on Placebo Maintenance (N=26) | All Treated Patients - Induction (N=157)
Abdomen, Pain (Gastrointestinal disorders) | 3 | 0 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 4 | 50
Anorexia (Metabolism and nutrition disorders) | 6 | 3 | 27
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5
Constipation (Gastrointestinal disorders) | 1 | 1 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 6
Creatinine increased (Investigations) | 3 | 0 | 6
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 15 | 3 | 44
Dizziness (Nervous system disorders) | 3 | 1 | 5
Dry Mouth (Gastrointestinal disorders) | 3 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 11
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5
Edema, head and neck (General disorders) | 2 | 1 | 1
Edema, limb (General disorders) | 2 | 0 | 9
Fatigue (General disorders) | 10 | 10 | 53
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 23
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3 | 5
Hypertension (Vascular disorders) | 2 | 2 | 7
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0 | 13
Joint pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 6
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 9
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3 | 1 | 27
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
Nausea (Gastrointestinal disorders) | 7 | 4 | 50
Neuropathy, sensory (Nervous system disorders) | 5 | 3 | 22
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 9
Platelet count decreased (Investigations) | 0 | 0 | 12
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 | 5 | 25
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 | 1 | 4
Rigors/chills (General disorders) | 2 | 1 | 2
Taste disturbance (Nervous system disorders) | 2 | 0 | 14
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0 | 8
Vomiting (Gastrointestinal disorders) | 3 | 0 | 22
Weight loss (Investigations) | 2 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less